CLINICAL TRIAL: NCT05805085
Title: Clinical Evaluation of Biomedics 1 Day Toric and MyDay Toric
Brief Title: Clinical Evaluation of Hydrogel and Silicone Hydrogel Daily Disposable Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-146
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-03

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (Experimental): Participants wore Lens A for 15 minutes (Period 1)
  Interventions: Device: Lens A
- Lens B (Experimental): Participants wore Lens B for 15 minutes (Period 2)
  Interventions: Device: Lens B

INTERVENTIONS:
Device: Lens A — Hydrogel Daily Disposable Toric Contact Lens for 15 minutes
  Arms: Lens A
Device: Lens B — Silicone Hydrogel Daily Disposable Toric Contact Lens for 15 minutes
  Arms: Lens B

SUMMARY:
This study was to evaluate the patient subjective experiences of two daily disposable toric contact lenses.

DETAILED DESCRIPTION:
This was a participant masked, interventional, prospective, direct refit, bilateral wear study. The purpose of this study was to evaluate the patient subjective experiences of a hydrogel daily disposable toric contact lens when compared to a silicone hydrogel daily disposable toric contact lens after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

A person was eligible for inclusion in the study if he/she:

* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and signed an information consent letter.
* Self-reports having a full eye examination in the previous two years.
* Anticipates being able to wear the study lenses for at least 8 hours a day, 5 days a week.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Habitual soft contact lens wearers who currently wear toric contact lenses, or use spectacles for all distances vision correction, for the past 3 months minimum.
* Has a contact lens spherical prescription between plano to - 10.00 (inclusive) best corrected visual acuity of 20/30 or better in either eye.
* Has refractive astigmatism no less than -0.75D and no more than 1.75D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease.
* Has read, understood, and signed the information consent letter.

Exclusion Criteria:

A person was excluded from the study if he/she:

1. Is participating in any concurrent clinical or research study.
2. Has any known active ocular disease and/or infection that contraindicates contact lens wear.
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable.
4. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable.
5. Has known sensitivity to the diagnostic sodium fluorescein used in the study.
6. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment.
7. Has undergone refractive error surgery or intraocular surgery.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan G Carracedo Rodríguez, OD, MSc, PhD, Principal Investigator — University Complutense of Madrid
Locations (1):
- Clinic of Optometry; Faculty of Optics and Optometry, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens A: All participants wore Lens A for 15 minutes (Period 1)
- Lens B: All participants wore Lens B for 15 minutes (Period 2)
Period: Period 1: Lens A, 15 Minutes
Arm/Group | Lens A | Lens B
Started | 40 | 0 (All participants received Lens A in Period 1.)
Completed | 40 | 0
Not Completed | 0 | 0
Period: Period 2: Lens B, 15 Minutes
Arm/Group | Lens A | Lens B
Started | 0 (All participants received Lens B in Period 2.) | 40
Completed | 0 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes study participants that completed all study visits
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was stratified by sex (Male and Female)
  years
    Male: number analyzed (Participants) | 13
    Male | 27.10 (6.04)
    Female: number analyzed (Participants) | 27
    Female | 27.08 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Handling at Insertion, Dispensing Visit
Description: Subjective handling an lens insertion was assessed at the dispending visit using a 0-100 scale, where 100=Excellent, very easy; 0=Very difficult to manage. Collected once at the end of 15 minutes of wear.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lens A: Participants that received Lens A
- Lens B: Participants that received Lens B
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 40 | 40
score on a scale | 87.13 (13.68) | 88.50 (10.14)

2. Primary Outcome: Subjecting Handling at Insertion, Follow-up Visit
Description: Subjective handling at lens insertion was assessed at the follow-up visit using a 0-100 scale, where 100=Excellent, very easy; 0=Very difficult to manage. Collected once at the end of 15 minutes of wear.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 40 | 40
score on a scale | 92.63 (9.28) | 90.13 (9.97)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 2 days
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT05805085/Prot_SAP_000.pdf